CLINICAL TRIAL: NCT00384787
Title: A Phase Ib Clinical Trial to Compare the Safety, Tolerability, and Immunogenicity of an HIV-1 Adenoviral Vector Boost Administered Intramuscularly, Intradermally, or Subcutaneously After an HIV-1 DNA Plasmid Vaccine Prime Administered Intramuscularly to Healthy Adenovirus Type 5 Seropositive HIV-1-Uninfected Adults
Brief Title: Safety of and Immune Response to a DNA HIV Vaccine Followed by an Adenoviral Vaccine Boost Given Three Different Ways to HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 069; 10391 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Adenoviral Vector Vaccine; DNA Plasmid Vaccine; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

ARMS (3):
- 1 (Experimental): Group 1 will receive three vaccinations with the HIV DNA vaccine. Vaccinations will be given at study entry and Months 1 and 2. Participants will also receive an adenoviral vaccine boost intramuscularly at Month 6.
  Interventions: Biological: VRC-HIVDNA009-00-VP; Biological: VRC-HIVADV014-00-VP
- 2 (Experimental): Group 2 will receive three vaccinations with the HIV DNA vaccine. Vaccinations will be given at study entry and Months 1 and 2. Participants will also receive an adenoviral vaccine boost intradermally at Month 6.
  Interventions: Biological: VRC-HIVDNA009-00-VP; Biological: VRC-HIVADV014-00-VP
- 3 (Experimental): Group 3 will receive three vaccinations with the HIV DNA vaccine. Vaccinations will be given at study entry and Months 1 and 2. Participants will also receive an adenoviral vaccine boost subcutaneously at Month 6.
  Interventions: Biological: VRC-HIVDNA009-00-VP; Biological: VRC-HIVADV014-00-VP

INTERVENTIONS:
Biological: VRC-HIVDNA009-00-VP — HIV DNA vaccine containing the HIV genes gag, pol, nef, and env A,B, and C. The HIV DNA vaccine will be given in three doses intramuscularly at study entry and Months 1 and 2
Biological: VRC-HIVADV014-00-VP — Adenoviral vector HIV booster vaccine containing the HIV genes gag, pol, and env. The adenoviral vector HIV booster vaccine will be administered intramuscularly (Group 1), intradermally (Group 2), or subcutaneously (Group 3) at Month 6

SUMMARY:
The purpose of this study is to determine the safety of, immune response to, and tolerability of an adenoviral vector HIV vaccine given after a three-dose regimen of a DNA HIV vaccine. The adenoviral vaccine will be given into arm muscle (intramuscularly), between skin layers (intradermally), or under the skin (subcutaneously).

NOTE: In October 2007, vaccinations with the adenoviral vaccine, VRC-HIVADV014-00-VP, were discontinued. In December 2007, vaccinations with the DNA vaccine were also discontinued. Participants will be followed for safety and immune responses at regular study visits.

DETAILED DESCRIPTION:
One factor that may affect safety and immunogenicity to an HIV vaccine is the route of vaccine administration. Administration into the skin (intradermal) or subcutaneous tissue may be more immunogenic or provide a different pattern of immune responses than administration by the intramuscular route. Previous studies with other preventive vaccines suggest that the resulting immunogenicity following intradermal or subcutaneous vaccine administration is comparable or better than immunogenicity observed following intramuscular administration. Increased immunogenicity though use of a particular route will likely result in greater demonstrated efficacy, requiring fewer or lower doses of vaccine to elicit a sufficient immune response.

The DNA HIV vaccine VRC-HIVDNA009-00-VP has shown immunogenicity in multiple clinical trials; in one trial, the DNA vaccine demonstrated a nearly 100% CD4 T-cell response rate. The adenoviral vector HIV vaccine VRC-HIVADV014-00-VP has shown immunogenicity when given intramuscularly and has appeared safe and well tolerated in prior vaccine trials in HIV uninfected adults. The DNA plasmids in both vaccines code for proteins from HIV subtypes A, B, and C. This study will evaluate the safety, immunogenicity, and tolerability to a DNA HIV vaccine, followed by an adenoviral vaccine boost given either intramuscularly, intradermally, or subcutaneously, in HIV uninfected adults.

All participants will receive three doses of the DNA vaccine intramuscularly at study entry and Months 1 and 2. Participants will be randomly assigned to one of three groups, differing by how they will receive the adenoviral vaccine boost:

* Group 1 participants will receive the vaccine boost intramuscularly at Month 6
* Group 2 participants will receive the vaccine boost intradermally at Month 6
* Group 3 participants will receive the vaccine boost subcutaneously at Month 6

This study will last 1 year. There will be 12 study visits; a physical exam, medication history, and risk reduction/pregnancy prevention compliance counseling will occur at all visits. Urine and blood collection will occur at selected visits. Participants will be asked to complete a social impact assessment at Months 2, 6, and 12 and an outside testing and belief questionnaire at Months 6 and 12. Participants will be asked to record their temperature and other side effects in a symptom log on the day of each vaccination and for 3 days thereafter to report any side effects.

NOTE: In October 2007, vaccinations with the adenoviral vaccine, VRC-HIVADV014-00-VP, were discontinued. In December 2007, vaccinations with the DNA vaccine were also discontinued. Participants will be followed for safety and immune responses at regular study visits and will be asked to continue in long term follow-up for purposes of safety surveillance to a total of 5 years following initial vaccination

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 and -2 uninfected
* Good general health
* Pre-existing adenovirus 5 (Ad5) neutralizing antibody titers of a 1:12 ratio or greater
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (anti-HCV) antibody negative or negative HCV PCR if anti-HCV antibody is positive
* Have access to a participating HIV Vaccine Trials Unit (HVTU) and are willing to be followed during the study
* Willing to receive HIV test results
* Able to understand the vaccination procedure
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV trial. Participants who can provide documentation that they received a placebo in a prior HIV trial may be eligible.
* Immunosuppressive medications within 168 days prior to first study vaccination
* Blood products within 120 days prior to first study vaccination
* Immunoglobulin within 60 days prior to first study vaccination
* Live attenuated vaccines within 30 days prior to first study vaccination
* Investigational research agents within 30 days prior to first study vaccination
* Medically indicated subunit or killed vaccines within 14 days prior to first study vaccination
* Allergy treatment with antigen injections within 30 days prior to first study vaccination
* Current anti-tuberculosis (TB) preventive therapy or treatment
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health. More information about this criterion can be found in the protocol.
* Any medical, psychiatric, or social condition that would interfere with the study. More information about this criterion can be found in the protocol.
* Any job-related responsibility that would interfere with the study
* Serious adverse reactions to vaccines, including hypersensitivity and related symptoms. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection. Participants who have been fully treated for syphilis more than 6 months prior to study entry are not excluded.
* Moderate to severe asthma. More information on this criterion can be found in the protocol.
* Type 1 or type 2 diabetes mellitus. Participants with histories of isolated gestational diabetes are not excluded.
* Thyroid disease or surgical removal of the thyroid requiring medication during the 12 months prior to study entry
* Accumulation of fluid in the blood vessels (angioedema) within 3 years prior to study entry if episodes are considered serious or have required medication in the 2 years prior to study entry
* Uncontrolled hypertension
* Body mass index (BMI) of 40 or greater OR BMI of 35 or greater if certain other criteria apply. More information about these criteria can be found in the protocol.
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that is unlikely to recur are not excluded.
* Seizure disorder
* Absence of the spleen
* Mental illness that would interfere with the study
* Pregnancy, breastfeeding, or plan to become pregnant during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse events) | After each injection and for 12 months after the first injection
Magnitude of HIV-specific T-cell responses assessed by the magnitude of IFN-gamma enzyme-linked immunosorbent spot (ELISpot) responses | 4 weeks after adenoviral vaccine boost

SECONDARY OUTCOMES:
Titer of HIV-specific binding antibodies assessed by enzyme-linked immunosorbent assay (ELISA) | 4 weeks after adenoviral vaccine boost

CONTACTS AND LOCATIONS:
Overall Officials: Beryl Koblin, PhD, Study Chair — New York Blood Center; Martin Casapia, MD, Study Chair — Asociación Civil Impacta Salud y Educación (IMPACTA), Peru
Locations (7):
- United States (6):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - NY Blood Ctr./Union Square CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- ACSA CRS, Iquitos, Maynas, Peru

REFERENCES:
- [Background] Barouch DH, Nabel GJ. Adenovirus vector-based vaccines for human immunodeficiency virus type 1. Hum Gene Ther. 2005 Feb;16(2):149-56. doi: 10.1089/hum.2005.16.149. PMID 15761255
- [Background] Kenney RT, Frech SA, Muenz LR, Villar CP, Glenn GM. Dose sparing with intradermal injection of influenza vaccine. N Engl J Med. 2004 Nov 25;351(22):2295-301. doi: 10.1056/NEJMoa043540. Epub 2004 Nov 3. PMID 15525714
- [Background] Pittman PR, Kim-Ahn G, Pifat DY, Coonan K, Gibbs P, Little S, Pace-Templeton JG, Myers R, Parker GW, Friedlander AM. Anthrax vaccine: immunogenicity and safety of a dose-reduction, route-change comparison study in humans. Vaccine. 2002 Jan 31;20(9-10):1412-20. doi: 10.1016/s0264-410x(01)00462-5. PMID 11818160
- [Background] Shiver JW, Emini EA. Recent advances in the development of HIV-1 vaccines using replication-incompetent adenovirus vectors. Annu Rev Med. 2004;55:355-72. doi: 10.1146/annurev.med.55.091902.104344. PMID 14746526
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067
- [Derived] Koblin BA, Casapia M, Morgan C, Qin L, Wang ZM, Defawe OD, Baden L, Goepfert P, Tomaras GD, Montefiori DC, McElrath MJ, Saavedra L, Lau CY, Graham BS; NIAID HIV Vaccine Trials Network. Safety and immunogenicity of an HIV adenoviral vector boost after DNA plasmid vaccine prime by route of administration: a randomized clinical trial. PLoS One. 2011;6(9):e24517. doi: 10.1371/journal.pone.0024517. Epub 2011 Sep 12. PMID 21931737